CLINICAL TRIAL: NCT00852124
Title: Safety of VSL#3 for Adult Asthmatics
Brief Title: Safety of VSL#3 in Adult Asthmatics
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Inadequate recruitment
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Mucosal Biology Research Center, Director Mucosal Biology Research Center, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HP-00040151; 1R21AT004089-01A1 (NIH)
Record Dates: First submitted 2009-02-13; First posted 2009-02-26 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2023-04-20 (Actual); Status verified 2022-11

CONDITIONS: Asthma
Keywords: Asthma; Probiotic; VSL#3
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Packets similar to VSL#3 will be taken 2 X daily but not containing active bacteria
  Interventions: Biological: VSL#3 or placebo
- VSL#3 (Active Comparator): Packets of VSL#3 (powder containing 8 bacteria believed to be beneficial) will be taken 2 x daily in food or a cool beverage.
  Interventions: Biological: VSL#3

INTERVENTIONS:
Biological: VSL#3 — VSL#3 2 times daily
  Arms: VSL#3
Biological: VSL#3 or placebo — 1 packet 2 x daily of placebo
  Arms: Placebo

SUMMARY:
We are proposing to test the safety of the probiotic, VSL#3, in a placebo controlled double blind safety study in 30 asthmatic adults. This adult safety trial was requested by the FDA IND review of a pediatric asthma protocol.

Adults with a doctor diagnosis of persistent asthma will take VSL#3 or placebo twice daily for 3 months. Data will be collected, including age, race, height, and weight, present medications, past medical history with emphasis on signs/symptoms of asthma.

On visits to the clinic we will evaluate

* Changes in lung function
* Intestinal permeability
* Intestinal bacteria
* Levels of inflammation in the blood
* Women will have repeat urine pregnancy testing at each clinic visit

DETAILED DESCRIPTION:
The monitored parameters that will be assessed at each clinic visit or phone call include:

1. the number of days with asthma related symptoms of cough, wheeze, dyspnea, awakening at night, and exercise limitation.
2. the number of asthma-related missed school/work days
3. the amount of use of asthma rescue medications
4. use of non-inhaled steroids
5. change in medications from baseline visit
6. diarrhea/liquid stools (> 2/day)
7. constipation
8. gas/bloating
9. fever/chills
10. scheduled or unscheduled visits for health care

To monitor for increased risk of safety concerns, we will also inquire on follow up visits and phone calls about the following:

1. household member with immunosuppression such as HIV or chemotherapy.

On visits to the clinic we will evaluate lung function by spirometry:

1. change in lung function with spirometry.
2. women of childbearing potential will have repeat urine pregnancy testing at each clinic visit.
3. intestinal barrier function
4. intestinal flora
5. serum inflammatory cytokines and IgE

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18-64 years old.
2. Doctor diagnosis of mild persistent asthma. Persistent asthma is defined by NAEPP guidelines as asthma symptoms (cough/wheeze/dyspnea/exercise limitation)of greater than 2 times/week daytime or greater than 2 times/month at night over the previous month but less than continual and less than 5 nights/week.
3. FEV1 greater than 60% predicted for age/gender/race/height based on normative data.
4. No unscheduled asthma related health visit in the 1 month prior to enrollment
5. School or work days missed less than or equal to 2 in the previous month for asthma.
6. Albuterol use less than 8 doses (2 puffs or one neb) in past week.
7. Ability to speak and understand English.
8. Telephone access.
9. Women of childbearing potential must confirm that they will use birth control while in the study and have a negative urine pregnancy screen at baseline.

Exclusion Criteria:

1. Pregnant women, prisoners.
2. Chronic illness (other than asthma, allergic rhinitis and eczema) such as renal disease, diabetes, hypertension or terminal disease or abnormal vital signs: T> 100.3F, HR>130 bpm, SBP>155 mmHg, or DBP>100 mmHg, RR>25 bpm, or pox<93% room air.
3. Unable to perform spirometry, necessary for lung function assessment.
4. Received probiotic in past 6 months.
5. Subject or household member has immunosuppression such as HIV, history of organ transplantation, present cancer or chemotherapy, primary immune disease, or is taking an immune modulating drug.
6. Severe persistent asthmatics who have continual daily or frequent (greater than 5 nights/week) asthma symptoms and/or FEV1 less than 60% predicted .
7. Diarrhea or constipation (symptoms more than once in the past week)
8. Unable to feed orally or to consume cornstarch
9. Lung disease other than asthma (e.g. COPD, cystic fibrosis, lung cancer, bronchiectasis, interstitial lung disease).
10. Subjects at increased risk of developing infective endocarditis such as those with a history of cardiac surgery, IV drug abuse, recent invasive medical procedures or dental work (recent = last month).
11. Allergy to Vancomycin or Cefepime. The parameters of intestinal barrier function, intestinal flora, serum inflammatory cytokines, IgE, will have no exclusion ranges as these will be collected over time on product as a way of describing the population characteristics of study participants.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2007-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessio Fasano, M. D., Principal Investigator — MBRC
Locations (1):
- University of Maryland Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Background] Bienenstock J, Wiley RE, Neigh GS, Waserman S, Keith P. Probiotics in the management and prevention of atopy. Clin Rev Allergy Immunol. 2002 Jun;22(3):275-85. doi: 10.1007/s12016-002-0012-z. No abstract available. PMID 12043385
- [Background] Hijazi N, Abalkhail B, Seaton A. Diet and childhood asthma in a society in transition: a study in urban and rural Saudi Arabia. Thorax. 2000 Sep;55(9):775-9. doi: 10.1136/thorax.55.9.775. PMID 10950897
- [Background] Kalliomaki M, Isolauri E. Role of intestinal flora in the development of allergy. Curr Opin Allergy Clin Immunol. 2003 Feb;3(1):15-20. doi: 10.1097/00130832-200302000-00003. PMID 12582309
- [Background] Bjorksten B, Naaber P, Sepp E, Mikelsaar M. The intestinal microflora in allergic Estonian and Swedish 2-year-old children. Clin Exp Allergy. 1999 Mar;29(3):342-6. doi: 10.1046/j.1365-2222.1999.00560.x. PMID 10202341
- [Background] Hijazi Z, Molla AM, Al-Habashi H, Muawad WM, Molla AM, Sharma PN. Intestinal permeability is increased in bronchial asthma. Arch Dis Child. 2004 Mar;89(3):227-9. doi: 10.1136/adc.2003.027680. PMID 14977697
- [Background] Isolauri E, Salminen S; Nutrition, Allergy, Mucosal Immunology, and Intestinal Microbiota (NAMI) Research Group Report. Probiotics: use in allergic disorders: a Nutrition, Allergy, Mucosal Immunology, and Intestinal Microbiota (NAMI) Research Group Report. J Clin Gastroenterol. 2008 Jul;42 Suppl 2:S91-6. doi: 10.1097/MCG.0b013e3181639a98. PMID 18542035
- [Background] Kalliomaki M, Salminen S, Poussa T, Isolauri E. Probiotics during the first 7 years of life: a cumulative risk reduction of eczema in a randomized, placebo-controlled trial. J Allergy Clin Immunol. 2007 Apr;119(4):1019-21. doi: 10.1016/j.jaci.2006.12.608. Epub 2007 Feb 7. No abstract available. PMID 17289135
- [Background] Laitinen K, Kalliomaki M, Poussa T, Lagstrom H, Isolauri E. Evaluation of diet and growth in children with and without atopic eczema: follow-up study from birth to 4 years. Br J Nutr. 2005 Oct;94(4):565-74. doi: 10.1079/bjn20051503. PMID 16197582
- [Background] Von Ehrenstein OS, Von Mutius E, Illi S, Baumann L, Bohm O, von Kries R. Reduced risk of hay fever and asthma among children of farmers. Clin Exp Allergy. 2000 Feb;30(2):187-93. doi: 10.1046/j.1365-2222.2000.00801.x. PMID 10651770
- [Background] Noverr MC, Noggle RM, Toews GB, Huffnagle GB. Role of antibiotics and fungal microbiota in driving pulmonary allergic responses. Infect Immun. 2004 Sep;72(9):4996-5003. doi: 10.1128/IAI.72.9.4996-5003.2004. PMID 15321991
- [Background] Kalliomaki M, Salminen S, Arvilommi H, Kero P, Koskinen P, Isolauri E. Probiotics in primary prevention of atopic disease: a randomised placebo-controlled trial. Lancet. 2001 Apr 7;357(9262):1076-9. doi: 10.1016/S0140-6736(00)04259-8. PMID 11297958
- [Background] Pessi T, Sutas Y, Hurme M, Isolauri E. Interleukin-10 generation in atopic children following oral Lactobacillus rhamnosus GG. Clin Exp Allergy. 2000 Dec;30(12):1804-8. doi: 10.1046/j.1365-2222.2000.00948.x. PMID 11122221
- [Background] Isolauri E, Sutas Y, Kankaanpaa P, Arvilommi H, Salminen S. Probiotics: effects on immunity. Am J Clin Nutr. 2001 Feb;73(2 Suppl):444S-450S. doi: 10.1093/ajcn/73.2.444s. PMID 11157355
- [Background] Weizman Z, Asli G, Alsheikh A. Effect of a probiotic infant formula on infections in child care centers: comparison of two probiotic agents. Pediatrics. 2005 Jan;115(1):5-9. doi: 10.1542/peds.2004-1815. PMID 15629974
- [Background] Land MH, Rouster-Stevens K, Woods CR, Cannon ML, Cnota J, Shetty AK. Lactobacillus sepsis associated with probiotic therapy. Pediatrics. 2005 Jan;115(1):178-81. doi: 10.1542/peds.2004-2137. PMID 15629999
- [Background] Cannon JP, Lee TA, Bolanos JT, Danziger LH. Pathogenic relevance of Lactobacillus: a retrospective review of over 200 cases. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):31-40. doi: 10.1007/s10096-004-1253-y. PMID 15599646
- [Background] Rinne M, Kalliomaki M, Arvilommi H, Salminen S, Isolauri E. Effect of probiotics and breastfeeding on the bifidobacterium and lactobacillus/enterococcus microbiota and humoral immune responses. J Pediatr. 2005 Aug;147(2):186-91. doi: 10.1016/j.jpeds.2005.03.053. PMID 16126047

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between December 2010 and November 2012. Participants were recruited via flyers and newsletters.
Groups:
- Placebo: Packets similar to VSL#3 taken 2 X daily but not containing active bacteria
  VSL#3 or placebo : 1 packet 2 x daily of placebo
- VSL#3: Packets of VSL#3 (powder containing 8 bacteria believed to be beneficial)taken 2 x daily in food or a cool beverage.
  VSL#3 : VSL#3 2 times daily
Period: Overall Study
Arm/Group | Placebo | VSL#3
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Zero participants analyzed for the primary outcome due to early termination of study
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | VSL#3 | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 3 |  | 3
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 3 |  | 3
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Safety of VSL#3 in Adults Asthmatics
Description: Change in FEV in adult asthmatics receiving VSL3# as compared to controls receiving placebo.
Time Frame: 3 months
Population: 3 people were randomized to placebo arm but no data were analyzed due to early termination of study and small number of patients enrolled.
Arm/Group | Placebo
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: No participants received Investigational Product. All thre particpants randomized to placebo arm. Recruitment was ended due to failure to recruit when PI relocated.
Arm/Group | Placebo | VSL#3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=3) | VSL#3 (N=0)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 3 (12) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Fever (Infections and infestations) | 1 (1) | 0 (0) — Associated with sinus infection
Sinus Infection (Infections and infestations) | 2 (2) | 0 (0)
Viral illness (Infections and infestations) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination due to small number of persons recruited before PI relocated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No